CLINICAL TRIAL: NCT04809363
Title: A Phase 4 Study Evaluating Real-World Use of CDPATH™, a Crohn's Disease Risk Prediction Tool
Brief Title: A Study of CDPATH™ to Help Manage and Treat Crohn's Disease
Acronym: COMPASS-CD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Vedolizumab-4015
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDPATH™ (Experimental): Participants with CD will be using CDPATH™ tool. Clinical data will be collected via an ongoing registry. Participants and health care provider (HCP)-reported outcomes data will be collected periodically once every 6 months for up to 36 months via electronic surveys. Two baseline blood samples will be collected at screening for CDPATH™ analysis. 1 additional sample will be collected for future potential biomarker analysis.
  Interventions: Other: CDPATH™; Other: Blood Draw

INTERVENTIONS:
Other: CDPATH™ — Crohn's disease risk prediction tool.
  Other Names: PROSPECT
Other: Blood Draw — Three blood samples will be drawn.

SUMMARY:
CDPATH™ is a tool to help predict the potential for developing Crohn's disease related complications in certain adult participants within 3 years. The main aim of the study is to explore the use of CDPATH™ to describe a participant's risk profile and to have discussions with their doctor about the potential path of their Crohn's disease. The number of visits will be decided by the study clinic according to their standard practice.

DETAILED DESCRIPTION:
The tool being tested in this study is called CDPATH™. CDPATH™ is being used to provide a graphical representation of an individual participant's risk of developing a CD-related complication within three years, leveraging known participant risk factors based on clinical, serologic and genetic variables to help people categorize risk who have CD. This study will gather data on the use of the tool in real-world settings to inform practical use of CDPATH™.

The study will enroll approximately 200 patients. Participants and health care providers (HCPs) will be surveyed to understand their satisfaction with the CDPATH™ process and with their treatment choice.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 36 months. Participants will make multiple visits to the HCP's clinic, and data will be collected approximately every six months up to 3 years, based on the timing of routine follow-up appointments for assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has an initial diagnosis of CD established within five years prior to screening by clinical and endoscopic evidence and corroborated by a histopathology report (if available).
2. Has agreed to use the CDPATH™ tool.
3. Has reliable access to the internet and is willing to answer electronic patient-reported outcomes (ePROs) throughout the study.

Exclusion Criteria:

1. Has had known complications from CD including but not limited to: bowel stricture, CD-related intra-abdominal abscess, internal penetrating disease (known fistula other than perianal fistula), non-perianal surgery, bowel resection, or stricturoplasty. A perianal fistula or abscess without other signs of penetrating disease is allowed.
2. Has had any non-CD-related abdominal surgery.
3. Has received investigational biologic or nonbiologic agents for the treatment of CD in an investigational protocol. Approved biologic or nonbiologic agents for CD are allowed.
4. Has previously used CDPATH™ or PROSPECT results to assess CD risk for complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Real-world Practice in Each Risk Category at Baseline Based on the CDPATH™ Tool Results | Baseline (Day 1)
  The risk profile of an individual participant with CD is the output of the CDPATH™ tool. Categories for CD includes low, medium, high risk of developing a CD complication within 3 years.

SECONDARY OUTCOMES:
Percentage of Participants with Specific Treatment Path and Choice Based on CDPATH™ Tool, Stratified According to Risk Category | Up to 36 months
  Treatment path (i.e., sequence over time) and choice, by low, medium and high risk, will be chosen to characterize treatment path and choice based on risk stratification.
Change From Baseline in Decisional Conflict Scale (DCS) Score | Baseline, then every 6 months up to 36 months
  DCS is a validated electronic patient-reported outcome (ePRO) collected via electronically administered patient surveys. It measures personal perceptions of the following responses: uncertainty in choosing options, modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making, and effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. DCS involves answering 11 questions of PRO, of which 10 questions can be answered as yes (score = 0) or unsure (score = 2) or no (score =4). The total score will range from 0 to 40. Higher score indicates higher decisional conflict.
Change From Baseline in Work Productivity and Activity Impairment Questionnaire - CD Version (WPAI-CD) Score | Baseline, then every 6 months up to 36 months
  WPAI-CD is a validated ePRO collected via electronically administered patient surveys. It consists of six questions that evaluate 4 domain scores: absenteeism (i.e., work time missed), presenteeism (i.e., reduced work productivity), overall work impairment, and activity impairment. Scores are expressed as a percentage of impairment, where higher scores indicate greater impairment and reduced productivity. The total score ranges from 0 (no impairment) to 100% (total loss of work productivity).
Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale Score | Baseline, then every 6 months up to 36 months
  PROMIS Global Health scale is a validated ePRO collected via electronically administered patient surveys. It is a 10-item PRO measuring the overall evaluation of one's physical and mental health. The total score ranges from 0 to 100. The final score will be represented by the T-score metric, in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. A higher PROMIS T-score represents more of the concept being measured (higher Global Health score indicate better health).
Patient-Reported Satisfaction and Experience Score with the CDPATH™ Tool | Up to 36 months
  Participant's satisfaction and experience with the CDPATH™ tool will be assessed based on 15 questions. Negative responses/lower score to/in these questions indicates less satisfaction whereas positive responses/higher score indicates satisfaction with the tool.
Number of Participants with Clinical Outcomes | Up to 36 months
  Participants with clinical outcomes describing the disease burden based on treatment path and controlling for risk strata will be reported.
Percentage of Participants with Healthcare Resource Utilization | Up to 36 months
  Healthcare resource includes healthcare provider (HCP) visits/referrals, visit to emergency room, hospitalizations, surgery, new CD-related complications, and diagnostic evaluations (e.g., imaging, colonoscopy, etc.).
Change from First Assessment in Health Care Provider (HCP)-reported Assessment of the Feasibility and Usability of the CDPATH™ Tool | First assessment (6 months after HCPs first enrolled participant) up to HCP leaves the study or the study ends (up to 36 months)
  HCP-reported CDPATH™ satisfaction data will be collected directly from HCPs via electronically administered HCP surveys and entered into the eCRF. HCPs will be queried regarding their satisfaction and experience with the general process, the ease of incorporating the tool in their everyday practice, and the impact of the tool on their treatment recommendations and participant communications. For the 6 questions, HCP will rate on 1-5 scale where, 1=strongly disagree and 5=strongly agree. For remaining 4 questions, written feedback from HCP will be consider. Overall positive responses will indicate higher feasibility and usability.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (44):
- United States (44):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, California
  - United Medical Doctors, Murrieta, California
  - University of Southern California Medical Center, Newport Beach, California
  - Clinnova Research Solutions, Orange, California
  - University of California at Irvine Medical Center, Orange, California
  - Kaiser Permanate of Colorado, Aurora, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Grand Teton Research Group, PLL, Idaho Falls, Idaho
  - GI Alliance, Arlington Heights, Illinois
  - GI Alliance, Gurnee, Illinois
  - Comprehensive Gastrointestinal Health, Northbrook, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Indiana University, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - GI Alliance - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Gastro Center of Maryland, Columbia, Maryland
  - Lahey Clinic Inc. - PARENT ACCOUNT, Burlington, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - Lenox Hill Hospital, New York, New York
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - The Oregon Clinic, P.C., Portland, Oregon
  - Susquehanna Research Group, LLC, Camp Hill, Pennsylvania
  - Allegheny Center for Digestive Health, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Palmetto Primary Care Physician Division of Gastroenterology, Summerville, South Carolina
  - Rapid City Medical Center, LLC, Rapid City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas at Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - GI Alliance - Southlake, Southlake, Texas
  - Care Access Research Berkley, Ogden, Utah
  - University of Utah, Salt Lake City, Utah
  - GCGA Physicians LLC, Fairfax, Virginia
  - Gastroenterology Associates, Lynchburg, Virginia
  - GI Alliance, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/605cd65feb9d7e001f5bc6a2